CLINICAL TRIAL: NCT02347098
Title: Plaque Regression and Progenitor Cell Mobilization With Intensive Lipid Elimination Regimen (PREMIER), Phase II
Acronym: PREMIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLIN-010-09S-1
Record Dates: First submitted 2015-01-20; First posted 2015-01-27 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Acute Coronary Artery Syndrome
Keywords: plaque; LDL; statin; endothelial; apheresis; acute coronary artery syndrome
MeSH Terms: conditions — Plaque, Amyloid | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- intensive LDL-lowering therapy (ILLT) (Experimental): Patient of acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) is randomized to LDL-apheresis and an oral daily dose of 40-80mg of Atorvastatin or equivalent.
  Interventions: Device: intensive LDL-lowering therapy; Drug: standard statin monotherapy
- standard statin monotherapy (SMT) (Active Comparator): Patient of acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) is randomized to an oral daily dose of 40-80mg of Atorvastatin or equivalent without LDL-apheresis
  Interventions: Drug: standard statin monotherapy

INTERVENTIONS:
Device: intensive LDL-lowering therapy — The intensive LDL-lowering therapy uses LDL-apheresis in addition to the standard statin therapy. The device used in this study is the LIPOSORBER LA-15 System, manufactured by Kaneka Pharma America LLC. A filter separates plasma from whole blood, the Liposorber -columns remove LDL from the plasma. The system recombines plasma and blood cells and returns them into the patient's body. This procedure typically takes about 3 hours. The procedure provides an immediate reduction in a patient's lipid levels. A single apheresis treatment can lower LDL by more than 80%, but levels return to baseline within 3 weeks.
  Other Names: LIPOSORBER LA-15 System
  Arms: intensive LDL-lowering therapy (ILLT)
Drug: standard statin monotherapy — The standard statin therapy of 40-80mg oral daily dose of Atorvastatin or other equivalent types of statin to lower LDL in blood for both randomized groups.
  Other Names: Atorvastatin or other equivalent types of statin

SUMMARY:
The purpose of this randomized, multi-site, clinical trial is to determine whether intensive therapy consisting of cholesterol-lowering statin drugs plus apheresis to cleanse the blood of low-density lipoprotein (LDL) cholesterol is more effective than statin therapy alone in reducing plaque volume in heart arteries of patients who have already suffered an acute coronary syndrome (ACS). The study will also investigate whether this intensive approach can help increase the presence of endothelial progenitor cells (EPC), stem cells that have been shown to reduce cardiovascular (CV) events in ACS patients. This study has two phases and FDA approval for phase II has been received and all information has been updated to reflect PREMIER Phase II.

DETAILED DESCRIPTION:
Using statins to lower blood cholesterol, and specifically LDL, is well established as a long-term strategy to reduce CVs and even death. But the most intensive pharmacologic lipid-lowering therapy with statins, though proven superior to standard dose regimens, is still associated with an unacceptably high rate of recurrent CV events early after an ACS. This study hypothesizes that for ACS patients undergoing percutaneous coronary intervention (PCI), intensive lipid-lowering therapy consisting of statins and LDL-apheresis (ILLT) will significantly reduce the total coronary atheroma volume of vulnerable plaque and augment mobilization of peripherally circulating EPC colony forming units, compared to guideline statin monotherapy (SMT). ILLT will lead to fewer CV events for these patients.

Patients presenting at four VA sites with ACS will be screened and consented before undergoing uncomplicated PCI (balloons or stents) and intravascular ultrasound with virtual histology (IVUS-HS). They will then be randomized into the ILLT arm or SMT arm of the study. The ILLT group will receive one treatment of LDL-apheresis plus a daily oral 40- 80mg dose of Atorvastatin or equivalent statin; the SMT group will only get 40-80mg Atorvastatin or equivalent. Patients will again undergo IVUS-HS 12 weeks after enrollment to measure atheroma volume; EPC level will also be checked.

The three-year duration of the study includes 24 months of accrual, six months of follow-up, and 12 months of study closure and data analysis. A two-sample t-test of mean difference with 90% power and 0.65 Cohen's D effect size provides a total sample size estimate of 102. Counting 20% drop-out rate, the sample size increases to 128.

The recent FDA recommendations regarding the design of the study have been included in the revised study protocol:

1. The safety data will be submitted to the FDA.
2. Patients will be randomized to both LDL-apheresis and an oral daily dose of 40-80mg Atorvastatin or equivalent statin (Intensive LDL-lowering therapy/ILLT) or a daily dose of 40-80mg of Atorvastatin or equivalent statin without LDL-apheresis (standard statin monotherapy/SMT) following an uncomplicated PCI.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent (including HIPAA)
* Age >30 years
* Presenting with acute coronary syndrome (ACS), manifested as unstable angina or non-ST-elevation myocardial infarction
* Referred for clinically-indicated, non-emergent (the procedure is not required to be performed within 3 hours after patient presentation) coronary angiography and PCI with Intravascular Ultrasound with Virtual Histology (IVUS-VH) of target coronary artery for ACS
* Successful placement of two large bore IV cannulas in bilateral upper extremities
* Fasting (12 hrs.) LDL 70mg/dl while on less than or equal to 80mg Atorvastatin or equivalent dose of other statin, performed at time of admission or prior to PCI.

Exclusion Criteria:

* Known allergy to aspirin, clopidogrel, statins, or iodinated contrast
* Positive pregnancy test, planning to become pregnant, or breast-feeding
* Coexisting conditions that limit life expectancy to less than six months or affect patient compliance
* Uncontrolled fasting (12 hrs.) triglyceride levels ( 500mg/dl)
* Already participating in an investigational device or drug study
* History of heparin induced thrombocytopenia (HIT)
* Persons with estimated glomerular filtration rate (eGFR) of less than 45 ml/min
* ST-elevation myocardial infarction at admission
* Abnormal liver function test (LFT) at time of admission or prior to PCI with abnormal LFT defined as any liver transaminases (ALT or AST) 3 times the upper limit of the normal laboratory reference
* Pre-PCI or post-PCI left ventricular ejection fraction <25% by echo or cardiac catheterization done after admission
* Pre-PCI, intra-PCI, or post-PCI hemodynamic instability with hypotension
* Pre-PCI, intra-PCI, or post-PCI cardiac arrest
* Pre-PCI or post-PCI acute heart failure with or without pulmonary edema
* Intra-PCI or post-PCI sustained ventricular tachycardia
* Complicated PCI, defined as PCI with any of the vascular access complications (large hematoma with lump > 5 cm or requiring medical treatment; arteriovenous (AV) fistula; pseudo aneurysm requiring treatment; retroperitoneal bleeding), or PCI with any of the procedural complications (abrupt vessel closure; no-reflow phenomenon; new angiographic thrombus; new major dissection with reduced flow; catheter-related thrombus), or PCI requiring further medical treatments (urgent coronary artery bypass graft (CABG); endotracheal intubation; unplanned in-aortic balloon pump; left ventricular assist device (LVAD); covered stent; unplanned temporary pacemaker wire; administration of inotropes; cardiopulmonary resuscitation (CPR)) , or PCI resulting in clinical events (death; stroke; myocardial infarction; stent thrombosis) during or within 24 hours after the index PCI
* Post-PCI ongoing chest pain
* Post-PCI severe groin pain and hematoma > 5cm in diameter
* Persons whose hemoglobin is less than 9 grams following the index PCI/IVUS procedure, or who experience a drop in hemoglobin of greater than or equal to 2 grams following the procedure
* Not able to comply with study protocol as determined by the investigators

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (4):
- United States (4):
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kole A, Hua F, Wei Y, Carlson K, Hayenga HN, Banerjee S. Analysis of Plaque Characteristics by Virtual Histology-Intravascular Ultrasound in Short-Term Follow-Up Post-Acute Coronary Syndrome and Association With Lipid-Lowering Therapy: Insights From the PREMIER Trial. J Am Heart Assoc. 2023 May 16;12(10):e028873. doi: 10.1161/JAHA.122.028873. Epub 2023 May 9. No abstract available. PMID 37158083
- [Derived] Banerjee S, Luo P, Reda DJ, Latif F, Hastings JL, Armstrong EJ, Bagai J, Abu-Fadel M, Baskar A, Kamath P, Lippe D, Wei Y, Scrymgeour A, Gleason TC, Brilakis ES. Plaque Regression and Endothelial Progenitor Cell Mobilization With Intensive Lipid Elimination Regimen (PREMIER). Circ Cardiovasc Interv. 2020 Aug;13(8):e008933. doi: 10.1161/CIRCINTERVENTIONS.119.008933. Epub 2020 Aug 14. PMID 32791950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment for Phase II pivotal study started on March 30, 2015, and the first participant was randomized on April 9, 2015. The recruitment period stopped in July 2017. For all 4 participating sites, Dallas, Nashville, Oklahoma City, and Denver randomized 80, 5, 38, and 6 participants, respectively.
Pre-assignment Details: There were 270 subjects consented and enrolled into the study before entering catheterization lab to have the PCI procedure, but 141 subjects were not randomized to treatment assignments with the major exclusion reason as not able to comply with study protocol based on the inclusion/exclusion criteria.
Groups:
- Intensive LDL-lowering Therapy (ILLT): Patient of acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI) is randomized to LDL-apheresis in addition to the standard statin therapy of an oral daily dose of 40-80mg of Atorvastatin or equivalent. The device used in this study is the LIPOSORBER LA-15 System, manufactured by Kaneka Pharma America LLC. A filter separates plasma from whole blood, the Liposorber -columns remove LDL from the plasma. The system recombines plasma and blood cells and returns them into the patient's body. This procedure typically takes about 3 hours. The procedure provides an immediate reduction in a patient's lipid levels. A single apheresis treatment can lower LDL by more than 80%, but levels return to baseline within 3 weeks.
Period: Overall Study
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Started | 63 | 66
Completed | 56 | 58
Not Completed | 7 | 8
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Refuse Follow-up Visit | 1 | 5
Not completed — no visit due to illness | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT) | Total
Number analyzed (Participants) | 63 | 66 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.4) | 67.3 (7.7) | 65.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 62 | 65 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 14 | 27
  White | 48 | 52 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 66 | 129
Weight [Mean (Standard Deviation); unit: pounds] | 225.0 (56.7) | 221.7 (46.7) | 223.3 (51.6)
Height [Mean (Standard Deviation); unit: inches] | 69.9 (2.7) | 70.0 (2.9) | 70.0 (2.8)
Heart Rate [Mean (Standard Deviation); unit: beats/min] | 79.0 (16.0) | 71.8 (13.6) | 75.3 (15.2)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 140.0 (22.1) | 141.8 (23.9) | 140.9 (22.9)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 78.7 (13.1) | 77.0 (13.1) | 77.8 (13.1)
Smoker [Count of Participants; unit: Participants]
  Never | 16 | 12 | 28
  Current | 16 | 14 | 30
  Former | 31 | 40 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in the Total Atheroma Volume From Baseline to 12 Weeks
Description: The primary effectiveness outcome measure was the change in the total atheroma volume within a ≥ 20 mm long segment of the target coronary artery from baseline to 12 weeks post-PCI. The measurement was done via IVUS-VH at 2 time points (baseline during index PCI and 90-day follow-up).
Time Frame: 12 weeks
Population: Reported results are based on observed data from participants who had primary outcome measured.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Number analyzed (Participants) | 56 | 58
mm^3 | -7.63 (23.78) | -3.10 (17.74)
Statistical Analysis 1: Comparison: Intensive LDL-lowering Therapy (ILLT) vs Standard Statin Monotherapy (SMT); Test type: Superiority; p = 0.2533, t-test, 2 sided

2. Secondary Outcome: Change in % Necrotic Core Component of Atheroma
Description: The %NC component of atheroma were obtained via IVUS-VH at 2 time points (baseline during index PCI and 90-day follow-up).
Time Frame: 12 weeks
Population: Reported results are based on observed data from participants who had secondary outcome measured.
Measure: Mean (Standard Deviation); unit: percentage of atheroma component
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Number analyzed (Participants) | 45 | 48
percentage of atheroma component | 0.44 (6.81) | 0.94 (9.89)
Statistical Analysis 1: Comparison: Intensive LDL-lowering Therapy (ILLT) vs Standard Statin Monotherapy (SMT); Test type: Superiority; p = 0.7790, t-test, 2 sided

3. Secondary Outcome: Endothelial Progenitor Cell Colony Forming Units/ml of Peripheral Blood Across Time
Description: The cell culture assay and quantification of circulating EPC-CFU were performed for patients recruited at the Dallas VA center only. The assay were done at 4 time points (pre-PCI, post-PCI, 30-day follow-up, and 90-day follow-up).
Time Frame: 12 weeks
Population: Reported results are based on observed data from participants who had secondary outcome measured. This outcome was captured for Dallas site only.
Measure: Mean (Standard Deviation); unit: colonies/ml
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Number analyzed (Participants) | 37 | 35
colonies/ml
  baseline pre-PCI | 11.85 (9.24) | 11.99 (11.37)
  baseline post-PCI | 15.30 (10.96) | 17.89 (16.91)
  30-day | 21.60 (14.78) | 20.40 (17.87)
  90-day | 16.32 (13.29) | 15.06 (14.33)
Statistical Analysis 1: Comparison: Intensive LDL-lowering Therapy (ILLT) vs Standard Statin Monotherapy (SMT); Test type: Superiority; p = 0.4549, Mixed Models Analysis — The p-value reported compares the trends of outcome across time (baseline pre-PCI, baseline post-PCI, 30-day follow-up, and 90-day follow-up) between treatment groups using the repeated measurement analysis

4. Secondary Outcome: Major Adverse CV Events
Description: The number of patients who experienced major adverse cardiovascular endpoints (MACE) including death, myocardial infarction, coronary revascularization, and stroke during the follow-up periods.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
Number analyzed (Participants) | 63 | 66
Participants | 5 | 2
Statistical Analysis 1: Comparison: Intensive LDL-lowering Therapy (ILLT) vs Standard Statin Monotherapy (SMT); Test type: Superiority; p = 0.2663, Fisher Exact

ADVERSE EVENTS:
Time Frame: AE/SAE/UADE were monitored at the study sites throughout the whole period of the study at each clinic visit and telephone contact, beginning as soon as a study participant signs the Informed Consent and continuing through end-of-study for each participant. Most participants were followed for around 6 months for AE/SAE/UADE.
Description: All AE/SAE/UADE including both those related to the study intervention and those not related to the intervention, will be collected and recorded on the appropriate case report forms (CRF). For the purpose of safety monitoring, the study intervention is defined as the use of 1) statins with or without the addition of LDL-apheresis, 2) LDL-apheresis, and 3) cardiac catheterization and IVUS-VH as described in this protocol.
Arm/Group | Intensive LDL-lowering Therapy (ILLT) | Standard Statin Monotherapy (SMT)
All-Cause Mortality (participants affected / at risk) | 2/63 | 0/66
Serious Adverse Events (participants affected / at risk) | 28/63 | 28/66
Other Adverse Events (participants affected / at risk) | 42/63 | 39/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive LDL-lowering Therapy (ILLT) (N=63) | Standard Statin Monotherapy (SMT) (N=66)
Coronary artery disease (Cardiac disorders) | 5 (5) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 7 (7)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 5 (5)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 5 (5) | 5 (5)
Vascular stent restenosis (General disorders) | 3 (3) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive LDL-lowering Therapy (ILLT) (N=63) | Standard Statin Monotherapy (SMT) (N=66)
Chest pain (General disorders) | 7 (7) | 6 (6)
Procedural hypotension (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 1 (1)
Flushing (Vascular disorders) | 6 (6) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 3 (3)
Renal cyst (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephropathy (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Our study is limited by its relatively small sample size and short follow-up. All study sites were Veterans Affairs medical centers and therefore enrolled a disproportionate number of men, limiting the generalizability of its findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT02347098/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT02347098/SAP_001.pdf